CLINICAL TRIAL: NCT05176314
Title: A Phase 1, Open-Label, Drug Interaction Study to Investigate the Effect of Single and Multiple Doses of Pirtobrutinib on the Pharmacokinetics of Rosuvastatin in Healthy Participants
Brief Title: A Drug Drug Interaction (DDI) Study of Pirtobrutinib (LY3527727) and Rosuvastatin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Loxo Oncology, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 18366; J2N-MC-JZNW (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-01-03; First posted 2022-01-04 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium; pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rosuvastatin + Pirtobrutinib (Experimental): Participants received study intervention through oral administration as follows:
  * Day 1: 20 milligram (mg) rosuvastatin alone
  * Day 6: 20 mg rosuvastatin co-administered with 200 mg pirtobrutinib
  * Days 7 to 12: Once daily (QD) doses of 200 mg pirtobrutinib alone
  * Day 13: 20 mg rosuvastatin co-administered with 200 mg pirtobrutinib
  * Days 14 to 17: QD doses of 200 mg pirtobrutinib alone.
  Interventions: Drug: Rosuvastatin; Drug: Pirtobrutinib

INTERVENTIONS:
Drug: Rosuvastatin — Administered Orally.
Drug: Pirtobrutinib — Administered Orally.
  Other Names: LY3527727

SUMMARY:
The main purpose of this study is to determine the effect of pirtobrutinib on the levels of rosuvastatin in the blood stream in healthy participants. This study will also evaluate the safety and tolerability of rosuvastatin when administered in combination with pirtobrutinib in healthy participants. This study will last up to approximately 26 days excluding screening period.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and vital signs.
* Body mass index (BMI) within the range of 18.0 to 32.0 kilograms per meter squared (kg/m²) and a body weight of at least 50 kg.
* Males, or female participants who are not of childbearing potential.

Exclusion Criteria:

* Have known allergies to pirtobrutinib or rosuvastatin, related compounds, or any components of the formulation.
* Have an abnormal blood pressure and/or pulse rate, deemed to be clinically significant by the investigator.
* Have a significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, neurological, or psychiatric disorder or surgery (including cholecystectomy) capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational product; or of interfering with the interpretation of data.
* Have used or intend to use prescription or nonprescription medication (including dietary supplements, vitamins, and/or herbal medications), or modulators of CYP3A4 or BCRP within 7 days prior to dosing, unless, in the opinion of the investigator and sponsor, the medication will not interfere with the study.
* Have c.34AA, c.421AA, or c.34GA/421CA genotypes of ABCG2 as determined through genotyping.
* Have c.521TC and c/521CC genotypes of SLCO1B1 as determined by genotyping.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - QPS Bio-Kinetic Clinical Applications, Springfield, Missouri
  - Covance Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rosuvastatin + Pirtobrutinib
Started | 32
Safety Population Day 1, Day 6 and Days 7-12 (All participants who received at least one dose of study drug for the specified period.) | 32
Safety Population Day 13, Days 14-17 (All participants who received at least one dose of study drug for the specified period. One participant discontinued from the study at day 8 and didn't receive rosuvastatin + pirtobrutinib on day 13, and pirtobrutinib once daily (QD) on days 14 to 17, thus only 31 participants were analyzed for safety for that period.) | 31
Completed | 28
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Arm/Group | Rosuvastatin + Pirtobrutinib
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 15
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Rosuvastatin
Description: PK: Cmax of Rosuvastatin
Time Frame: Day 1, Day 6 and Day 13: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120 hours (h) post-dose.
Population: All randomized participants who received at least one dose of rosuvastatin and had evaluable PK data for the respective days for this outcome analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Rosuvastatin + Pirtobrutinib
Number analyzed (Participants) | 31
nanograms per milliliter (ng/mL)
  Day 1 | 9.45 (56)
  Day 6 | 23.0 (51)
  Day 13: number analyzed (Participants) | 30
  Day 13 | 23.0 (49)

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-inf]) of Rosuvastatin
Description: PK: AUC(0-inf) of Rosuvastatin
Time Frame: Day 1, Day 6 and Day 13: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120 hours (h) post-dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter(ng*h/mL)
Arm/Group | Rosuvastatin + Pirtobrutinib
Number analyzed (Participants) | 31
nanograms*hours per milliliter(ng*h/mL)
  Day 1: number analyzed (Participants) | 30
  Day 1 | 88.2 (44)
  Day 6 | 189 (41)
  Day 13: number analyzed (Participants) | 30
  Day 13 | 207 (40)

ADVERSE EVENTS:
Time Frame: Baseline to end of follow-up (up to 24 days).
Description: All participants from the safety population.
Groups:
- 20 mg Rosuvastatin (Day 1): Participants received 20 milligram (mg) rosuvastatin alone on day 1 through oral administration.
- 20 mg Rosuvastatin + 200 mg Pirtobrutinib (Day 6): Participants received 20 mg rosuvastatin co-administered with 200 mg pirtobrutinib on day 6 through oral administration.
- 200 mg Pirtobrutinib QD (Days 7-12): Participants received once daily (QD) doses of 200 mg pirtobrutinib alone on days 7 to 12 through oral administration.
- 20 mg Rosuvastatin + 200 mg Pirtobrutinib (Day 13): Participants received 20 mg rosuvastatin co-administered with 200 mg pirtobrutinib on day 13 through oral administration.
- 200 mg Pirtobrutinib QD (Days 14-17): Participants received QD doses of 200 mg pirtobrutinib alone on days 14 to 17 through oral administration.
Arm/Group | 20 mg Rosuvastatin (Day 1) | 20 mg Rosuvastatin + 200 mg Pirtobrutinib (Day 6) | 200 mg Pirtobrutinib QD (Days 7-12) | 20 mg Rosuvastatin + 200 mg Pirtobrutinib (Day 13) | 200 mg Pirtobrutinib QD (Days 14-17)
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 3/32 | 1/32 | 3/32 | 0/31 | 1/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 mg Rosuvastatin (Day 1) (N=32) | 20 mg Rosuvastatin + 200 mg Pirtobrutinib (Day 6) (N=32) | 200 mg Pirtobrutinib QD (Days 7-12) (N=32) | 20 mg Rosuvastatin + 200 mg Pirtobrutinib (Day 13) (N=31) | 200 mg Pirtobrutinib QD (Days 14-17) (N=31)
Headache (Nervous system disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT05176314/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT05176314/SAP_001.pdf